CLINICAL TRIAL: NCT03111524
Title: The Classroom Communication Resource (CCR) Intervention to Change Grade 7 Peer's Attitudes Towards Children Who Stutter (CWS) in the Western Cape: A Protocol for a Cluster-Randomised Controlled Trial
Brief Title: The Classroom Communication Resource (CCR) Intervention to Change Grade 7 Peer's Attitudes Towards Children Who Stutter (CWS)
Acronym: CCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rizwana Mallick (Other)
Collaborators: University of Cape Town (Other); National Research Fund - South Africa (Unknown)
Responsible Party: Sponsor-Investigator, Rizwana Mallick, PhD student; investigator, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PhD protocol 2017
Record Dates: First submitted 2017-03-09; First posted 2017-04-13 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Stuttering in Adolescence; Bullying of Child
Keywords: stuttering; children who stutter; peer attitudes; classroom-based intervention; teasing; bullying
MeSH Terms: conditions — Stuttering; Bullying

STUDY DESIGN:
Intervention Model Description: 10 schools are included. The schools are assigned to control versus intervention groups
Who Masked: Participant, Investigator
Masking Description: The Principal investigator is blinded to the study. The researcher is able to observe while the research assistants are aware of who is in the control versus intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Intervention school 1 (Active Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is administered by the teacher. The participants observe the intervention which is a social story (read by the teacher), the class performs a role-play (same plot as the story) and then the teacher facilitates and leads a semi-structured discussion. The intervention takes place in 1 classroom lesson only. No further intervention is completed.
  Interventions: Other: Classroom Communication Resource
- Intervention school 2 (Active Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is administered by the teacher.The participants observe the intervention which is a social story (read by the teacher), the class performs a role-play (same plot as the story) and then the teacher facilitates and leads a semi-structured discussion. The intervention takes place in 1 classroom lesson only. No further intervention is completed.
  Interventions: Other: Classroom Communication Resource
- Intervention school 3 (Active Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is administered by the teacher. The participants observe the intervention which is a social story (read by the teacher), the class performs a role-play (same plot as the story) and then the teacher facilitates and leads a semi-structured discussion. The intervention takes place in 1 classroom lesson only. No further intervention is completed.
  Interventions: Other: Classroom Communication Resource
- Intervention school 4 (Active Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is administered by the teacher. The participants observe the intervention which is a social story (read by the teacher), the class performs a role-play (same plot as the story) and then the teacher facilitates and leads a semi-structured discussion. The intervention takes place in 1 classroom lesson only. No further intervention is completed.
  Interventions: Other: Classroom Communication Resource
- Intervention school 5 (Active Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is administered by the teacher. The participants observe the intervention which is a social story (read by the teacher), the class performs a role-play (same plot as the story) and then the teacher facilitates and leads a semi-structured discussion. The intervention takes place in 1 classroom lesson only. No further intervention is completed.
  Interventions: Other: Classroom Communication Resource
- control school 1 (Placebo Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is not administered by the teacher.
  Interventions: Other: No intervention
- control school 2 (Placebo Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is not administered by the teacher.
  Interventions: Other: No intervention
- control school 3 (Placebo Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is not administered by the teacher.
  Interventions: Other: No intervention
- control school 4 (Placebo Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is not administered by the teacher.
  Interventions: Other: No intervention
- control school 5 (Placebo Comparator): All participants complete the questionnaire at baseline. The Classroom Communication Resource Intervention is not administered by the teacher.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Classroom Communication Resource — The Classroom Communication Resource intervention is a classroom- and group-based interventions administered by teachers. It includes a social story, role-play and teacher-led discussion
  Arms: Intervention school 1; Intervention school 2; Intervention school 3; Intervention school 4; Intervention school 5
Other: No intervention — No intervention is administered in this group as these are control groups
  Arms: control school 1; control school 2; control school 3; control school 4; control school 5

SUMMARY:
Children who stutter (CWS) are at high risk of being teased and bullied in primary school because of the negative peer attitudes and perceptions towards stuttering. Their experiences can lead to long-term negative psychosocial consequences which can in turn affect academic performance. There is little evidence to determine if classroom-based interventions are effective in changing peer attitudes to stuttering. This study is designed to assess whether a classroom-based CCR intervention versus usual practice in schools will lead to positive shift in attitudes about stuttering at 6-months among grade 7 students.

DETAILED DESCRIPTION:
Children who stutter (CWS) are placed at risk for being teased and bullied in Primary school (Blood & Blood, 2004; Blood, Boyle, Blood & Nalesnik, 2010; Evans, Healy, Kawai & Rowland, 2008; Langevin, Kleitman, Packman & Onslow, 2009) due to negative peer attitudes and perceptions (Blood & Blood, 2004; Blood et al., 2010; Evans at al., 2008; Langevin et al., 2009). Negative attitudes and interactions result in CWS being viewed as different or disabled leading to social rejection (Evans et al., 2008). Social rejection may lead to long term negative consequences such as reduced academic and social interactions, depression, and negative self-perceptions (Ferguson, Miguel, Kilburn & Sanchez, 2007; Hawker & Boulton, 2000) and are harmful if not urgently addressed. This is prevalent in the adolescent population due to stress and rapid changes of emotion at this age (Evans et al, 2008). Attitudes and perceptions overlap (Foster, 2006) which is useful as negative peer attitudes may lead to negative perceptions towards CWS (Blood & Blood, 2004; Blood et al., 2010; Evans et al., 2008; Langevin et al., 2009). While the relationships between attitudes, attitude change and behaviour change are complex and multifaceted (Prochaska, Redding & Evers 2008), this study focusseson f attitude as the precursor for change. (Scott, 2000). This study does not focus on behaviour change. Attitudes are described as an individual's evaluation of issues, objects and other individuals. The evaluation of another person or object can be positive or negative (Petty, Wegener & Tormala, 2003) Furthermore, attitude formation is known to continuously change over time, (Krahe & Altwasser, 2006) as it is learnt and shaped (Foster, 2006).

The International Classification and Functioning of Disability (ICF) framework (Murphy, Yaruss & Quesal., 2007) considers holistic management of the CWS. It advocates for classroom-based interventions to reduce teasing and bullying (Merrell, Gueldner , Ross & Isava., 2008; Murphy et al., 2007; Langevin, 2009) because children spend a large amount of time with teachers (Blank et al, 2009). Classroom-based interventions also empowers teachers. International public education addresses stuttering-related stigma (Scott, 2000) through reducing the debilitating nature of stuttering and improving social environments and reactions (St Louis, 2011). These publicised campaigns have not documented effectiveness. However, the potential for classroom-based interventions to change attitudes to stuttering are emerging. Survey of Human Attributes- Stuttering (POSHA-S) showed that negative attitudes are prevalent in school-aged children (Flynn & St Louis, 2011) A follow-up study conducted in South Africa, using the POSHA-S, showed that teachers were requesting assistance with managing negative attitudes to stuttering (Abrahams, 2015). The Teasing and Bullying: Unacceptable Behaviour (TAB) included teacher administered activities and yielded positive results pre- and post- intervention (; Langevin, 2009; Langevin & Prasad, 2012). The TAB was however not suitable for South African classrooms due to time and technology constraints as well as contextual, cultural and linguistic differences. This led to the development of the South African specific intervention, the CCR intervention. It was developed and has been refined since 2009 as part of a series of the University of Cape Town projects. The CCR intervention yielded positive results at 1 month post-intervention within the lower and higher quintile population respectively (Kathard et al.,2014 & Walters, 2015) and more so at 6 months post-intervention (Badroodien, 2015). The feasibility study thus reported potential effectiveness of the CCR intervention at 1 and 6 months post-intervention (Badroodien, 2015). The findings were however inconclusive as it called for a more rigorous design method. The findings also reported that a RCT was feasible despite concerns regarding the retention of participants. A RCT was thus recommended as the next stage in these projects (Badroodien, 2015) The CCR intervention addresses prosocial behaviours and skills, including but not limited to the promotion of positive behaviour change, peer support and resilience through intervention (Blank et al, 2009) in the areas of Positive Social Distance (PSD), Verbal Interaction (VI) and Social Pressure (SP) in the CCR intervention. The areas of PSD, VI and SP are additionally measured where PSD represents the overall ease, acceptance of and comfort a child feels when around CWS (Langevin, 2009; e.g. 'I would let a child who stutters hang out with us'). VI evaluates peer's negative thoughts, emotions and feelings, e.g. frustration experienced towards a CWS (Langevin et al., 2009). SP evaluates general thoughts regarding CWS through examining social pressure and subjective norms (Langevin, 2009). An example is 'I would be ashamed to be seen with a child who stutters'. The promotion of these prosocial behaviours and skills may facilitate the prevention of anxiety and depression (Blank et al, 2009). In post-apartheid schools are unequal particularly in relation to resources. IN an attempt to address such inequality, a system based on the National Norms and Standards for school funding policy was developed to classify schools in relation to resources..) . (Motala, 2006) using the National Norms and Standards for School Funding (NNSSF) policy (Mestry & Ndhlovu, 2014). Lower quintiles one, two and three are no fee paying schools (Department of Education, 2009; Sayed & Motala, 2012).Higher quintiles four and five are fee-paying schools that are better resourced (Department of Education, 2009; Sayed & Motala, 2012). This study therefore aims to compare the treatment effect in the low and high quintiles, explored as a subgroup in this study

ELIGIBILITY:
Inclusion Criteria:

Eligible participants for the primary objective of this study include grade 7 mixed- gender participants aged 11 and older attending public schools within the Cape Metro urban area across the lower (two and three) and higher (four and five) quintiles where the Language of learning and teaching (LoLT) is English.

Exclusion Criteria:

Participants in private schools, in grades 1-6 within the Cape Metro urban area with a LoLT other than English .

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Baseline rating of peer attitudes | Baseline
  The Stuttering Resource Outcomes Measure is used to evaluate peer's rating of attitudes towards children who stutter.
6 months post-intervention rating of peer attitudes | 6 months post-intervention
  The Stuttering Resource Outcomes Measure is used to evaluate peer's rating of attitudes towards children who stutter

SECONDARY OUTCOMES:
Construct peer ratings of attitudes | Baseline and 6 months post-intervention
  The Stuttering Resource Outcomes Measure is used to evaluate peer's rating of attitudes towards children who stutter. This questionnaire is made up of and measures the constructs: positive social distance, verbal interaction and social pressure. These constructs will be analsyed within constructs and compared to one another at each time frame

CONTACTS AND LOCATIONS:
Overall Officials: Lehana Thabane, Study Chair — McMaster University

IPD SHARING:
Plan to Share IPD: No
The individual participant data willl be shared amongst the primary researcher, research assistants, contributing authors and the statistician. Once the data is analysed, the findings will be reported in an article. The study looks at clusters and thus it is not necessary to share IPD. If any researchers are wanting access to statistical data, this can be requested

REFERENCES:
- [Derived] Borhan S, Mallick R, Pillay M, Kathard H, Thabane L. Sensitivity of methods for analyzing continuous outcome from stratified cluster randomized trials - an empirical comparison study. Contemp Clin Trials Commun. 2019 Jul 5;15:100405. doi: 10.1016/j.conctc.2019.100405. eCollection 2019 Sep. PMID 31338480
- [Derived] Mallick R, Kathard H, Borhan ASM, Pillay M, Thabane L. A cluster randomised trial of a classroom communication resource program to change peer attitudes towards children who stutter among grade 7 students. Trials. 2018 Nov 29;19(1):664. doi: 10.1186/s13063-018-3043-3. PMID 30497490
- [Derived] Mallick R, Kathard H, Thabane L, Pillay M. The Classroom Communication Resource (CCR) intervention to change peer's attitudes towards children who stutter (CWS): study protocol for a randomised controlled trial. Trials. 2018 Jan 17;19(1):43. doi: 10.1186/s13063-017-2365-x. PMID 29343283